CLINICAL TRIAL: NCT05387512
Title: Efficacy, Safety, and Cost-effectiveness Evaluation of the β2-Adrenergic Receptor Blocker ICI118551 Combined With a PD-1 Inhibitor in Patients With Non-Small Cell Lung Cancer
Brief Title: A Real World Study of β2-Adrenergic Blocker Plus PD-1 Inhibitor in Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Affiliated Hospital of Nantong University (Other)
Collaborators: The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-K002-01
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer
Keywords: lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Camrelizumab treatment group: Patients receive camrelizumab (an anti-PD-1 antibody) alone. Reference regimen of Camrelizumab 200mg/3 weeks will follow the approved product label or study protocol. This arm corresponds to the "ICB therapy" group in the foundational preclinical study.
  Interventions: Drug: Camrelizumab
- Camrelizumab + β-blocker Combination treatment group: Patients receive camrelizumab in combination with a β2-adrenergic receptor blocker (e.g., a selective agent such as ICI-118551 used in preclinical models, or a clinically available alternative like propranolol). The specific β-blocker, dosing, and schedule will be defined in the study protocol. This arm directly tests the translational hypothesis derived from the preclinical finding that β-blockade reverses T cell exhaustion and restores sensitivity to anti-PD-1 therapy.
  Interventions: Drug: β-adrenergic receptor blocker; Drug: Camrelizumab

INTERVENTIONS:
Drug: β-adrenergic receptor blocker — A β-blocker (specifically targeting the β2-adrenergic receptor, such as the selective antagonist ICI-118551 used in preclinical models, or a clinically available agent like propranolol) will be administered in combination with Camrelizumab. The specific agent, dose, route (e.g., oral), and schedule will be defined in the study protocol.
  Groups: Camrelizumab + β-blocker Combination treatment group
Drug: Camrelizumab — Camrelizumab is a humanized anti-PD-1 monoclonal antibody. The intervention will be administered as an intravenous infusion at a dose of 200 mg every 3 weeks, in accordance with the approved product label or the study protocol.
  Other Names: SHR-1210

SUMMARY:
This study aims to explore an optimized treatment regimen of camrelizumab for Chinese patients with non-squamous non-small cell lung cancer. We will evaluate the efficacy, safety, and cost-effectiveness of camrelizumab monotherapy versus camrelizumab combined with a beta-adrenergic receptor blocker. Based on real-world data, a Markov model will be established to analyze the incremental cost-effectiveness of the combination therapy compared to monotherapy. Deterministic sensitivity analysis and probabilistic sensitivity analysis will be performed.

DETAILED DESCRIPTION:
1. Evaluate the feasibility, safety, and preliminary efficacy of adding a β-adrenergic receptor blocker to standard anti-PD-1 immunotherapy (camrelizumab). Studies suggest that sympathetic nervous system signaling, mediated through β-adrenergic receptors on T cells, may contribute to T cell dysfunction and resistance to immune checkpoint inhibitors. Our aim is to pharmacologically inhibit this pathway to assess whether the functional capacity of tumor-infiltrating T cells can be modulated, thereby potentially restoring or enhancing sensitivity to camrelizumab. We will systematically monitor patient outcomes, including tumor response and progression-free survival, and compare them against benchmarks.
2. Concurrently, this study incorporates a comprehensive pharmacoeconomic analysis. The goal is to determine the cost-effectiveness of the combination strategy (camrelizumab plus β-blocker) compared to camrelizumab monotherapy within the Chinese healthcare context. This evaluation will be conducted using a decision-analytic Markov model, which simulates the long-term clinical trajectory and associated costs of patients under each treatment strategy. The model will be populated with efficacy and safety data generated from this study, supplemented by real-world data on resource utilization and costs. To assess the robustness of the economic conclusions, deterministic sensitivity analysis (examining the impact of varying key parameters) and probabilistic sensitivity analysis (incorporating uncertainty across all parameters) will be performed. This analysis aims to provide evidence regarding the value of the combination strategy to inform clinical practice and healthcare resource allocation decisions.

ELIGIBILITY:
Inclusion Criteria:

(1)Histologically confirmed advanced (stage IIIB/IV) NSCLC; (2) Planned to receive first-line anti-PD-1/L1 monotherapy and deemed suitable for such treatment; (3) Older than 18 years of age; (4) ECOG (Eastern Oncology Collaboration group) score 0-1; (5) Ecg and liver and kidney function are normal; (6) No second primary tumor disease or serious complications.

Exclusion Criteria:

(1) Known hypersensitivity to camrelizumab or any of its excipients, or to any component of the planned β-blocker; (2) Clear contraindications to the use of a β-adrenergic receptor blocker; (3)Active infection requiring systemic therapy;(4)Any other concurrent severe illness or clinical condition that, in the investigator's judgment, would interfere with the completion or interpretation of the study protocol or increase patient risk.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, pathological records and follow-up information of newly treated lung cancer patients in our hospital and four hospitals in Nanjing and Nantong from June 2022 to May 2025 were collected. Patients meeting the criteria of admission were divided into experimental group and control group.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 2022-2025
  Time from randomization until first documented disease progression per RECIST v1.1 (based on CT scans) or death from any cause. Tumor assessments by CT will be performed every 12 weeks (approximately every 3 cycles) during the first year, and annually thereafter until progression. The Kaplan-Meier method will be used to estimate the median PFS and its 95% confidence interval for each group, and survival curves will be plotted. Intergroup comparisons will be performed using the log-rank test. Additionally, a Cox proportional hazards model will be constructed to estimate the hazard ratio and its 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyuan Tang, Doctor, Study Director — Affilication Hospital of Nantong University
Locations (1):
- Department of Pharmacy, Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided